CLINICAL TRIAL: NCT06542510
Title: The Impact of Working Night Shifts on Cardiac Autonomic Nervous Regulation During the Six-minute Walk Test in Nurses
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-064
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Autonomic Nervous System Imbalance
Keywords: heart rate variability; night shift; autonomic nervous system; six-minute walk test; nurses
MeSH Terms: interventions — Shift Work Schedule

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: working night shift — working night shift
  Other Names: night shift

SUMMARY:
To evaluate changes in heart rate variability (HRV) after the six-minute walk test (6MWT) in nurses following a night shift and explore the impact of night shift work on the regulation of the autonomic nervous system in the heart.

Thirty-five female nurses, with a mean age of 28.7 years (range 21.0-37.0 years), participated in this study. On the first and second mornings after a night shift, the nurses performed the 6MWT. During the test, electrocardiogram (ECG) signals, blood pressure, and walking distance were recorded simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Female nurses aged ≥ 18 years who had undergone annual physical examinations, did not have serious cardiopulmonary diseases, and were able to walk normally were considered for inclusion in the study.

Exclusion Criteria:

* (ⅰ) having children at home who require night care; (ⅱ) current pregnancy; (ⅲ) engaging in activities that significantly impact heart rate, such as sexual activity, 24 hours before and 24 hours after working night shifts; (ⅳ) history of thyroid dysfunction, hypertension, diabetes, coronary heart disease, etc.; (ⅴ) experiencing upper respiratory tract infection, fever, cough, diarrhea, or other illnesses within 1 week before the planned enrollment; (ⅵ) consuming coffee or strong tea, smoking, drinking alcohol, or using other substances that affect heart rate 3 days before the planned enrollment; (ⅶ) taking β-receptor blockers, sleeping pills, psychotropic drugs, or other medications that affect heart rate; and (ⅷ) judged by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patient self-report
Study Population: The participants were nurses from Nanfang Hospital of Southern Medical University who worked ward shifts. The nurses in this study had one night shift every 5-10 days, from 00:00 a.m. to 8:00 a.m., followed by 2-3 days off.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Delta HRV during the 6MWT | 18 minutes
  On the first and second mornings after a night shift, the nurses performed the 6MWT.During the test, electrocardiogram (ECG) signals was recorded simultaneously.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data of the study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Zhan T, Wei X, Zhang Z, Shi Z, Xie H, Ma X, Pan S, Zha D. The impact of working night shifts on cardiac autonomic nervous regulation during the six-minute walk test in nurses. BMC Nurs. 2024 Dec 18;23(1):907. doi: 10.1186/s12912-024-02563-y. PMID 39696211